CLINICAL TRIAL: NCT02447211
Title: Topical Doxepin for Prevention and Management of Radiation-induced Dermatitis
Brief Title: Topical Doxepin for Radiation-induced Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Golnaz Vaseghi, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 900
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxepin cream (Active Comparator): Patients use doxepin cream 5% twice daily for two weeks
  Interventions: Drug: Doxepin cream 5%
- Placebo (Placebo Comparator): Patients use cream without doxepin ingredient twice daily for two weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxepin cream 5% — Patients use doxepin creamtwice daily for one weeks
  Arms: doxepin cream
Other: Placebo — Patients use cream without doxepin ingredient twice daily for one weeks
  Arms: Placebo

SUMMARY:
Radiation dermatitis is one of the most common side effects of radiotherapy approximately occurring in about 95% of patients receiving radiotherapy . Acute injury due to structural tissue damage, generation of free radicals, irreversible double-stranded breaks in nuclear and mitochondrial DNA, and initiation of an inflammatory response in the epidermis and dermis occurs within hours to weeks after radiation exposure. Radiation dermatitis due to pain and discomfort has an adverse impact on the quality of a patient's life.The radiation toxicities such as radiation dermatitis encountered in clinical practice are typically managed with a variety of topical agents such as water-based moisturizing creams or lotions, topical steroids, antiinflammatory emulsions, and wound dressings. Pharmacologic interventions for the prevention and treatment of these toxicity can be used to protect skin against radiation damage.Currently, there is no standard treatment for the prevention of radiation-induced dermatitis with demonstrated effectiveness.The aim of this randomized, double-blind, placebo-controlled study is to evaluate the effectiveness of topical doxepin for the prevention and management of radiation-induced dermatitis during postoperative radiotherapy for breast cancer.

DETAILED DESCRIPTION:
The patients who have undergone breast surgery and require radiotherapy and fulfill the inclusion criteria of the study will be entered the study. All the patients will be treated by 3D conformal radiation therapy using CT -based treatment planning and multi leaf linear accelerators. The patients will be treated by conventional fractionation regimens to a total dose of 5000 cGy (25 fractions of 200 cGy, 5 days per week). Every week the patients will be visited by an experienced radiation oncologist and the skin reaction will be determined and recorded according to RTOG Acute Radiation Morbidity Scoring Criteria which scores from 0 to 4. The patients receive Doxepin cream at the beginning of 5th week of radiotherapy and use it for a whole week. After acquiring written permission, the radiotherapy site will be photographed at the start and ending of the Doxepin

ELIGIBILITY:
Inclusion Criteria:

* Female with a diagnosis of, breast adenocarcinoma and be referred for post-operative radiotherapy with or without concurrent chemotherapy and with or without mastectomy
* Participants must not be pregnant.
* Participants treated with a total dose of 5000 cGy (25 fractions of 200 cGy, 5 days per week

Exclusion Criteria:

* Patients who are not eligible
* The presence of skin diseases in the radiation area
* Patients have constipation, xerostomia, blurred vision, urinary retention
* Hypersensitivity to doxepin

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Grading of dermatitis was performed according to the Radiation Therapy Oncology Group acute radiation morbidity scoring criteria | At the beginning of 5th week of radiotherapy to two weeks
  at the beginning of 5th week of radiotherapy and use it for two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Golnaz Vaseghi, Ph.D, Principal Investigator — Applied Physiology Research Center, Cardiovascular Research Institute, Isfahan University of Medical Sciences, Isfahan, Iran; Alireza Amouheidari, MD, Principal Investigator — Head, Department of Radiation Oncology,Isfahan Milad Hospital, Isfahan,Iran; Laleh Shariati, Ph.D, Principal Investigator — Isfahan University of Medical Sciences; Shaghayegh Shaghayegh Haghjoo-Javanmard, Ph.D, Study Director — Applied Physiology Research Center, Isfahan University of Medical Sciences, Isfahan, Iran; Hajar Naji, M.S, Study Chair — Applied Physiology Research Center, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran